CLINICAL TRIAL: NCT02589067
Title: Decolonization of the Oropharynx, an Important and Neglected Reservoir of S. Aureus Colonization.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 30529
Record Dates: First submitted 2015-10-20; First posted 2015-10-28 (Estimated); Results first posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-06

CONDITIONS: S. Aureus Oropharyngeal Colonization
MeSH Terms: interventions — chlorhexidine gluconate; Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Randomized to 15mL 0.12% Chlorhexidine Gluconate oral rinse, to be used twice daily for 60 seconds for 7 days.
  Interventions: Drug: Chlorhexidine gluconate
- Placebo (Placebo Comparator): Randomized to 15mL saline placebo oral rinse, to be used twice daily for 60 seconds for 7 days.
  Interventions: Drug: Saline Placebo

INTERVENTIONS:
Drug: Chlorhexidine gluconate — Oral rinse of either 0.12% Chlorhexidine Gluconate oral rinse to test the safety/efficacy of 0.12% Chlorhexidine Gluconate oral rinse in decolonizing the oropharynx of children colonized with S. aureus.
  Other Names: Peridex; Periogard
  Arms: Experimental
Drug: Saline Placebo — Placebo saline oral rinse to to test the safety/efficacy of 0.12% Chlorhexidine Gluconate oral rinse in decolonizing the oropharynx of children colonized with S. aureus.
  Arms: Placebo

SUMMARY:
The problem of interest is the high rate of recurrent SSTIs in children caused by S. aureus despite the use of systemic antibiotic treatment, due to difficulties in decolonization and the prevalence of antibiotic-resistant strains such as MRSA.

This problem will be studied through a randomized, double-blind, placebo-controlled clinical trial of the use of a 0.12% clorhexidine gluconate (CHG) oral rinse in decolonizing S. aureus in the oropharynx in children 5-17 years old. CHG is an excellent candidate for use in children as its safety has been widely established, and it is readily commercially available. Eligible, consented subjects will be asked to participate in a baseline study visit in which swabs of their oropharynx and nares are obtained, and they are educated on the use of either CHG oral rinse or a placebo oral rinse containing saline. The subjects will be instructed to perform the oral rinse twice daily for seven days. Two follow-up visits will occur at 7 and 28 days post-baseline, where subjects' nares and oropharynx are again swabbed in order to ascertain short- and long-term decolonization of S. aureus. This procedure will serve to 1) determine the efficacy of a CHG oral rinse in decolonization of S. aureus, 2) investigate the safety, tolerability, and compliance of oropharyngeal decolonization among children and their caregivers, and 3) determine the genetic backgrounds of strains of S. aureus associated with continued colonization.

DETAILED DESCRIPTION:
Each year, children visit doctors offices and emergency rooms over 2 million times due to skin and soft tissue infections (SSTIs). These SSTIs are usually caused by a bacteria called Staphylococcus aureus (S. aureus), and can result in severe negative consequences such as hospitalization, disability, and even death. Despite treatment with antibiotics, 20-70% of children with an SSTI will develop a recurrent infection within the next year. Additionally, this treatment fails to eradicate S. aureus from children nearly 50% of the time. Of the types of S. aureus that cause these infections, antibiotic-resistant strains such as methicillin-resistant S. aureus (MRSA), which are associated with higher rates of transmission, have become increasingly more common. Thus, the problem of interest is the high rate of recurrent SSTIs in children caused by S. aureus despite the use of systemic antibiotic treatment, due to difficulties in decolonization and the prevalence of antibiotic-resistant strains such as MRSA.

ELIGIBILITY:
Inclusion Criteria:

1. History of skin or soft tissue infection that occurred between 1 month and 5 years ago, regardless of whether antibiotics were given, as per patient report
2. Age > 5 years and < 18 years.
3. Able to gargle as assessed by verbal question.
4. Willing and able to undergo nares and oropharyngeal swabbing.
5. Able to come to the research clinic for study follow-up visits for the study period.

Exclusion Criteria:

1. Current suspected or confirmed infection requiring systemic antibiotics.
2. Receipt of systemic antibiotics in the prior 28 days.
3. Plans for administration or likely receipt of systemic antibiotics in the next 28 days (e.g., if the patient suffers from recurrent infections such as otitis media or has a planned surgery that requires prophylactic antibiotics).
4. Plans for hospitalization or likely hospitalization in the next 28 days (e.g., if the patient suffers from recurrent infections)
5. Any of the following in the prior 6 months: hemodialysis, peritoneal dialysis, central venous catheter placement, and systemic chemotherapy for cancer, any immune-compromising condition.
6. Previous participation in the study.
7. Pregnancy (all female subjects of childbearing age will be given a pregnancy test prior to enrollment).

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 67 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loren G Miller, MD, MPH, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (1):
- Los Angeles BioMedical Research Institute (LA BioMed), Torrance, California, United States

IPD SHARING:
Plan to Share IPD: Yes
After publication of trial results, data will be shared with investigators upon request to the Principal Investigator and after signing a Data Use Agreement.
Supporting Information: Study Protocol, SAP

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.12% Chlorhexidine Gluconate Oral Rinse: Randomized to 15mL 0.12% Chlorhexidine Gluconate oral rinse, to be used twice daily for 60 seconds for 7 days.
  Chlorhexidine gluconate: Oral rinse of either 0.12% Chlorhexidine Gluconate oral rinse to test the safety/efficacy of 0.12% Chlorhexidine Gluconate oral rinse in decolonizing the oropharynx of children colonized with S. aureus.
- Saline Placebo Oral Rinse: Randomized to 15mL saline placebo oral rinse, to be used twice daily for 60 seconds for 7 days.
  Saline Placebo: Placebo saline oral rinse to to test the safety/efficacy of 0.12% Chlorhexidine Gluconate oral rinse in decolonizing the oropharynx of children colonized with S. aureus.
Period: Overall Study
Arm/Group | 0.12% Chlorhexidine Gluconate Oral Rinse | Saline Placebo Oral Rinse
Started | 33 | 34
Completed | 28 | 28
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.12% Chlorhexidine Gluconate Oral Rinse | Saline Placebo Oral Rinse | Total
Number analyzed (Participants) | 33 | 34 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 33 | 34 | 67
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 11 (11.7) | 12.4 (11.7) | 11 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 19 | 21 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Hispanic | 29 | 29 | 58
  White Not Hispanic | 0 | 1 | 1
  Asian/Pacific Islander | 1 | 2 | 3
  Black/African American | 3 | 1 | 4
  other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 33 | 34 | 67

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Eradiction of S. Aureus From the Oropharyngeal at 7 Days
Description: The primary endpoint is eradication of S. aureus oropharyngeal colonization at 7 days using an intention to treat (ITT) model.
  .
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | 0.12% Chlorhexidine Gluconate Oral Rinse | Saline Placebo Oral Rinse
Number analyzed (Participants) | 33 | 34
Participants | 18 | 7

2. Secondary Outcome: Number of Participants Eradication of S. Aureus Oropharyngeal Colonization at 28 Days
Description: Secondary outcome is eradication of S. aureus oropharyngeal colonization at 28 days using an intention to treat (ITT) model.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | 0.12% Chlorhexidine Gluconate Oral Rinse | Saline Placebo Oral Rinse
Number analyzed (Participants) | 33 | 34
Participants | 13 | 5

3. Secondary Outcome: Number of Participants With Persistent Same Strain of S. Aureus Genetic Backgrounds at 28 Days
Description: We characterized isolates associated with breakthrough of oropharyngeal colonization. Here we show the breakthrough isolates of the same strain at 28 days.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Groups:
- Saline Placebo Oral Rinse,: Randomized to 15mL saline placebo oral rinse, to be used twice daily for 60 seconds for 7 days.
  Saline Placebo: Placebo saline oral rinse to to test the safety/efficacy of 0.12% Chlorhexidine Gluconate oral rinse in decolonizing the oropharynx of children colonized with S. aureus.
Arm/Group | 0.12% Chlorhexidine Gluconate Oral Rinse | Saline Placebo Oral Rinse,
Number analyzed (Participants) | 33 | 34
Participants | 4 | 11

4. Secondary Outcome: Number of Participants With Persistent Different Strain of S. Aureus Genetic Backgrounds at 28 Days
Description: We characterized isolates associated with breakthrough of oropharyngeal colonization. Here we show the breakthrough isolates of different strains at 28 days.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | 0.12% Chlorhexidine Gluconate Oral Rinse | Saline Placebo Oral Rinse,
Number analyzed (Participants) | 33 | 34
Participants | 4 | 7

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | 0.12% Chlorhexidine Gluconate Oral Rinse | Saline Placebo Oral Rinse
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/34
Other Adverse Events (participants affected / at risk) | 1/33 | 1/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.12% Chlorhexidine Gluconate Oral Rinse (N=33) | Saline Placebo Oral Rinse (N=34)
other (Gastrointestinal disorders) | 1 (1) | 1 (1) — Patient experienced vomiting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT02589067/Prot_SAP_000.pdf